CLINICAL TRIAL: NCT00239707
Title: Effect of GIP / GIP Analog in Type 2 Diabetes After a Meal
Brief Title: GIP: Glucose-dependent Insulinotropic Peptide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AG0056
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: insulin sensitivity; blood sugar
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Gastric Inhibitory Polypeptide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infusion 1 (Experimental): Normal Saline
  Interventions: Drug: GIP
- Infusion 2 (Placebo Comparator): GIP or modified GIP
  Interventions: Drug: Modified GIP
- Infusion 3 (Placebo Comparator): GIP or modified GIP, opposite of Infusion 2
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: GIP — One-time 20 ng/kg/min infusion over 3 hours
  Other Names: Glucose dependent insulinotropic peptide
  Arms: Infusion 1
Drug: Modified GIP — One-time infusion over 3 hours; dose to maintain desired biological effect of below 140 mg/dl
  Other Names: GIP analog
  Arms: Infusion 2
Drug: Normal Saline — one-time infusion over 3 hours
  Other Names: Saline
  Arms: Infusion 3

SUMMARY:
The purpose of this study is to test the safety of glucose-dependent insulinotropic peptide (GIP)/GIP Analog on people with Type 2 Diabetes.

DETAILED DESCRIPTION:
The small bowel makes a hormone called glucose-dependent insulinotropic peptide (GIP). It is released into the blood stream and goes to the pancreas. It works there with nutrients, especially glucose, in the digested food so that insulin is released in sufficient amounts from the pancreas. The insulin causes the nutrients from the food to be stored in the liver, fat and muscle until they are needed to provide energy. GIP also slows emptying of food from the stomach, which decreases the rate with which fats in food are broken down and stored. Once it is released into the blood, GIP is quickly broken down and becomes inactive. Individuals with type 2 diabetes do not make enough GIP and pharmacological doses of naturally occurring GIP do not increase insulin secretion in patients with type 2 diabetes. This study is testing a modified GIP (it had one amino acid difference from naturally occurring human GIP) that is not broken down as quickly in individuals with type 2 diabetes, to determine if it will improve insulin secretion, after eating, in patients with type 2 diabetes. The study will also compare its effects to that of naturally occurring, human GIP. Both human GIP and the modified GIP (GIP analog) are manufactured by peptide synthesis techniques (not extracted from human gut and not recombinant technology).

A screening visit will be performed including blood work, EKG and physical exam. If eligible, patients would be scheduled for three infusion visits 2 months apart, where they will receive a normal saline infusion on the first visit and GIP or GIP analog on the remaining visits. The infusion visits will begin approximately 6:45 a.m. and patients will have frequent blood sampling through an intravenous line over a period of 7 hours. An additional intravenous line will be placed for the infusion of either the normal saline, GIP or GIP analog over a period of 3 hours. Patients will be given a breakfast meal consisting of 550 calories (one egg, piece of toast with margarine, corn flakes 2% milk and a banana). They will be given 2 Extra-Strength Tylenol to determine time frame that food is emptied from stomach by measuring Tylenol levels in the blood. At the end of each study visit, patients will be given lunch, intravenous lines will be discontinued and they will be discharged to home.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Healthy Type 2 Diabetics
* Agree to stay off glucosidases for 3 days prior to infusion visits (Examples: Precose, Glyset)
* Agree to stay off Sulfonylureas 5 days prior to infusion visits (Examples: Glucotrol, Amaryl, glyburide, metformin
* Able to ingest 1000 mg Tylenol on study visits
* Able to consume study breakfast consisting of scrambled egg, white toast with margarine, corn flakes, 2% milk, banana at each infusion visit
* Female participants must have Hct > 36
* Male participant must have Hct > 38
* No kidney or liver disease per history and evidenced by blood and urine tests
* Physical Exam and EKG that do not contraindicate patient to be in the study

Exclusion Criteria:

* Taking the following medications: Insulin, or Thiazolidinediones, i.e. Avandia, Actos
* Pregnancy
* Steroid use within the past 3 months
* Recent infection, fever or chills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
GIP, glucose, insulin measured frequently during infusions | baseline, 2 months, and 4 months

SECONDARY OUTCOMES:
GLP-1, ghrelin measured frequently during infusions | baseline, 2 months, and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Egan, MD, Principal Investigator — Chief, Diabetes Section, National Institute on Aging
Locations (1):
- National Institute on Aging, Clinical Research Branch, Baltimore, Maryland, United States

REFERENCES:
- [Background] Elahi D, Andersen DK, Brown JC, Debas HT, Hershcopf RJ, Raizes GS, Tobin JD, Andres R. Pancreatic alpha- and beta-cell responses to GIP infusion in normal man. Am J Physiol. 1979 Aug;237(2):E185-91. doi: 10.1152/ajpendo.1979.237.2.E185. No abstract available. PMID 464094
- [Background] Nauck MA, Heimesaat MM, Orskov C, Holst JJ, Ebert R, Creutzfeldt W. Preserved incretin activity of glucagon-like peptide 1 [7-36 amide] but not of synthetic human gastric inhibitory polypeptide in patients with type-2 diabetes mellitus. J Clin Invest. 1993 Jan;91(1):301-7. doi: 10.1172/JCI116186. PMID 8423228
- [Background] Elahi D, McAloon-Dyke M, Fukagawa NK, Meneilly GS, Sclater AL, Minaker KL, Habener JF, Andersen DK. The insulinotropic actions of glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1 (7-37) in normal and diabetic subjects. Regul Pept. 1994 Apr 14;51(1):63-74. doi: 10.1016/0167-0115(94)90136-8. PMID 8036284
- [Derived] Chia CW, Odetunde JO, Kim W, Carlson OD, Ferrucci L, Egan JM. GIP contributes to islet trihormonal abnormalities in type 2 diabetes. J Clin Endocrinol Metab. 2014 Jul;99(7):2477-85. doi: 10.1210/jc.2013-3994. Epub 2014 Apr 8. PMID 24712564